CLINICAL TRIAL: NCT05934565
Title: Mindful Steps: Coupling Technology and Mind-Body Exercise to Facilitate Physical Activity in Chronic Cardiopulmonary Disease
Brief Title: Mindful Steps 2.0: Promoting Physical Activity in Patients With COPD and HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Brigham and Women's Hospital (Other); VA Boston Healthcare System (U.S. Federal Agency); University of Michigan (Other)
Responsible Party: Principal Investigator, Gloria Y. Yeh, Director of Mind-Body Research, BIDMC General Medicine Division; Associate Professor of Medicine, Harvard Medical School, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AT012166-01A1 (NIH)
Record Dates: First submitted 2023-06-22; First posted 2023-07-07 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Heart Failure
Keywords: Mind-Body Exercise; FitBit; Mindful Steps
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: 2-arm parallel remotely delivered randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Testing will be facilitated by study staff who are blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Steps (Experimental): Multi-modal web intervention including: pedometer with individualized step-count goals, motivational and educational content, online community forum, mind-body videos (short themed clips that support walking, plus library of mind-body exercises), online group mind-body exercise classes, star incentive system; educational booklet
  Interventions: Behavioral: Mindful Steps
- Usual Care (No Intervention): Pragmatic usual care (standard care through participant's healthcare provider including pharmacological treatment and general advice for physical activity); educational booklet

INTERVENTIONS:
Behavioral: Mindful Steps — Integrated website, activity tracker, and mind-body training
  Arms: Mindful Steps

SUMMARY:
The goal of this fully-remote randomized controlled trial is to test the efficacy of Mindful Steps in facilitating physical activity compared to usual standard of care among 136 patients with COPD and/or HF. The main question it aims to answer is can this intervention promote physical activity as measured by daily step counts in sedentary patients with COPD and/or HF. Participants will be randomized (1:1 ratio) to receive either the Mindful Steps intervention or usual care for 12 months, with both arms receiving a Walking for Health education booklet.

DETAILED DESCRIPTION:
This is a 2-arm parallel remotely delivered RCT. A total of 136 participants with COPD and/or HF will be randomized in a 1:1 ratio to one of 2 arms in a pragmatic design: 1) Mindful Steps multi-modal intervention, or 2) usual care (including an education booklet on walking). Subjects will participate in the intervention for 12 months. Testing will occur at baseline, 3, 6, 12 (end intervention), and 15 months (post-intervention follow up) for all participants. Physical activity as measured by pedometer (i.e., daily step counts) at 12 months is the primary outcome to assess the efficacy of the Mindful Steps intervention. Secondary outcomes include cognitive-behavioral measures that may relate to behavior change in a conceptual model (self-efficacy, intrinsic motivation, mindful awareness/interoception) as well as patient-centered clinical outcomes (HRQL, dyspnea, fatigue, PA engagement, sedentary behavior).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD (defined as cigarette smoking history > 10 pack-years, and either a ratio of FEV1 to forced vital capacity < 0.70 or chest CT evidence of emphysema) OR clinical diagnosis of HF syndrome (with left ventricular systolic dysfunction or preserved ejection fraction and New York Heart Association Class 1-3)
* Medical clearance from provider to participate in an exercise program
* Have an active email account; access to a computer device (desktop, laptop, tablet, or smartphone that supports the Fitbit app).

Exclusion Criteria:

* COPD or HF exacerbation in the previous month
* Inability to ambulate
* Inability to collect at least 7 of 14 days of baseline step counts
* Current participation in a cardiac or pulmonary rehabilitation program

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity | baseline, months 3, 6, 12, and 15
  Daily step counts will be measured as an objective proxy for physical activity using FitBit pedometers (FitBit Inspire 3)

SECONDARY OUTCOMES:
Change in self-efficacy | baseline, months 3, 6, 12, and 15
  Exercise self-efficacy will be measured using the Self-Efficacy for Exercise Scale and the Self-Efficacy for Managing Chronic Disease Scale. The Self-Efficacy for Exercise Scale a 9-item validated scale; scores range from 9-28, with a higher score meaning more self-efficacy. The Self-Efficacy for Managing Chronic Disease Scale is a 6-item visual analog scale; scores range from 1-10, with a higher score indicating higher self-efficacy.
Change in intrinsic motivation | baseline, months 3, 6, 12, and 15
  Intrinsic motivation will be measured using the Intrinsic Motivation Inventory. This is a 22-item scale validated with four sub-scales: interest/enjoyment, perceived competence, perceived choice, and pressure/tension. A higher score is better, with a scoring range of 22-154.
Qualitative inquiry | months 6 and 12
  Half-hour semi-structured qualitative interviews guided by study staff will be conducted over video/phone in a random subset of 50 participants at the 6 and 12 month timepoints.
Change in disease-specific quality-of-life | baseline, months 3, 6, 12, and 15
  Disease-specific quality-of-life will be measured using St. George's Respiratory Questionnaire (SGRQ) and The Minnesota Living with Heart Failure Questionnaire (MLFHQ). The SGRQ is a 50-item instrument developed and validated in COPD and calculates four scores: symptomatology, activity, impacts and an overall metric; scores range from 0-100, with higher scores indicating more limitations. The MLFHQ is a 21-item instrument; total scores range from 0-105, with higher scores indicating poorer quality-of-life.
Change in exercise engagement | baseline, months 3, 6, 12, and 15
  Exercise engagement will be measured using the Community Healthy Activities Model Program for Seniors (CHAMPS) Physical Activity Questionnaire. This 41-item self-report questionnaire assesses engagement with physical activity, including frequency and duration, among older adults over the past 4 weeks. Separate scores are derived for physical activities of varying intensities. Frequency and estimated caloric expenditure are calculated per week for each of these physical activity categories, with higher scores indicating greater frequency and duration of exercise.
Change in sedentary behaviors/time | baseline, months 3, 6, 12, and 15
  Sedentary behaviors/time will be measured using online weekly exercise logs. These online weekly exercise logs will be used to assess frequency and categorize exercises.
Change in dyspnea | baseline, months 3, 6, 12, and 15
  Dyspnea is being measured using the UCSD Shortness of Breath Questionnaire - a 24 item questionnaire using a 6 point Likert scale; scores range from 0-120, with higher scores indicating greater dyspnea.
Change in fatigue | baseline, months 3, 6, 12 and 15
  Fatigue will be measured using the The Patient-Reported Outcome Measurement Information System (PROMIS) Fatigue Short Form 7a. Raw scores range from 7-35, and each raw score is translated into a standardized T-score, with higher T-scores representing greater fatigue.
Change in mindful awareness | baseline, months 3, 6, 12 and 15
  Mindful awareness will be measures using the Multidimensional Assessment of Interoceptive Awareness, consisting of 37 items (8 domains), each domain scored as the average score on a 6-point Likert.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - VA Boston, Boston, Massachusetts
  - BIDMC, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No